CLINICAL TRIAL: NCT07310927
Title: Alginate vs Sucralfate for GERD Symptomatic Relief in Combination With PPIS
Brief Title: Alginate vs Sucralfate for GERD Symptomatic Relief
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CMH Lahore Medical College and Institute of Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 580/2024
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Alginates; alginate, aluminium hydroxide, magnesium trisilicate, sodium bicarbonate drug combination; Sucralfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alginate Group (Experimental): Patient meeting the eligibility criteria will be given two tablespoons before meal twice a day along with PPIS.
  Interventions: Drug: Alginate
- Sucralfate Group (Active Comparator): Patient meeting the eligibility criteria will be given two tablespoons before meal twice a day along with PPIS.
  Interventions: Drug: Sucralfate

INTERVENTIONS:
Drug: Alginate — 2 Table spoon spoon suspension syrup twice a day before meal.
  Other Names: Gaviscon
  Arms: Alginate Group
Drug: Sucralfate — 2 Table spoon spoon suspension syrup twice a day before meal.
  Other Names: Ulsanic
  Arms: Sucralfate Group

SUMMARY:
Gastroesophageal reflux disease (GERD) is a chronic gastrointestinal disorder characterized by the regurgitation of gastric contents into the esophagus.It can also present in an atypical manner such as chest pain, dental erosions, chronic cough, laryngitis, or asthma i.e. extra gastroesophageal symptoms. Sucralfate is a unique anti-ulcer drug and is a basic aluminum salt of sucrose octa-sulfate. It forms a protective layer, enhancing bicarbonate production, demonstrating anti-peptic properties, and fostering tissue growth, regeneration, and repair and it undergoes minimal enteral reabsorption. Alginate is a naturally occurring anionic polymer typically obtained from brown seaweed and has been extensively investigated and used for many biomedical applications, due to its biocompatibility, low toxicity, relatively low cost, and mild gelation by addition of divalent cations such as Ca2+.Both sucralfate and alginate have been in use for the treatment and symptomatic relief of GERD and are well tolerated oral formulations.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) is a chronic gastrointestinal disorder characterized by the regurgitation of gastric contents into the esophagus. It is one of the most commonly diagnosed digestive disorders in the young adult population with a prevalence of 20%. Clinically GERD typically manifests with symptoms of heartburn and regurgitation. It can also present in an atypical manner such as chest pain, dental erosions, chronic cough, laryngitis, or asthma i.e. extra gastroesophageal symptoms. Several causative factors have been identified and implicated in the pathogenesis of GERD, like motor abnormalities such as esophageal dysmotility clearance, decrease tone of the lower esophageal sphincter (LES), transient LES relaxation, and delayed gastric emptying, and others are anatomical defects like hiatus hernia and obesity Sucralfate is a unique anti-ulcer drug and is a basic aluminum salt of sucrose octa-sulfate. It forms a protective layer, enhancing bicarbonate production, demonstrating anti-peptic properties, and fostering tissue growth, regeneration, and repair and it undergoes minimal enteral reabsorption. Alginate is a naturally occurring anionic polymer typically obtained from brown seaweed and has been extensively investigated and used for many biomedical applications, due to its biocompatibility, low toxicity, relatively low cost, and mild gelation by addition of divalent cations such as Ca2+.Alginate reacts with gastric acid, forming a gel-like raft that floats on the stomach contents. The raft acts as a physical barrier, preventing acid from reaching the esophagus. Both sucralfate and alginate have been in use for the treatment and symptomatic relief of GERD and are well tolerated oral formulations. This randomized clinical trial will oversee the effects of alginates versus sucralfate for GERD symptomatic relief in combination with proton pump inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* All patients having symptoms of severe GERD for more than 3 times /week

Exclusion Criteria:

1. Patients with preexisting cardiovascular disorders
2. Patients with chronic kidney or liver diseases
3. Patients with gross abnormalities on upper GI endoscopies e.g.; ulcers, tumors or those with history of upper GI surgery
4. Pregnant and breast feeding
5. Absence of Erosive esophagitis
6. Patients with peptic esophageal ulcers
7. PPI use within 4 weeks

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-29 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Reflux and Dyspepsia | Before Treatment, At 4 weeks, At 6 Weeks
  This involves questionnaire related to the symptoms and impact on quality of life.
  The total score is 140, ranging from 0 to 140, the higher the score the worse will be the symptoms.

SECONDARY OUTCOMES:
Adverse Effects and Tolerability | Before Treatment, At 2 weeks, At 4 Weeks
  Using Structured AE Forms and A 5-Point Tolerability Scale
Gerd Symptom Severity | Before Treatment, At 2 weeks, At 4 Weeks
  Using the 0-4 GERD Symptom Severity Scale, total number of items 20. Total score is 80, ranging from 0 to 80, the higher the score the worse will be the symptoms.
Quality of Life (QOLRAD) | Before Treatment, At 2 weeks, At 4 Weeks
  Using The Validated 0-4-Point Likert QOLRAD Questionnaire, total number of items is 15.Total score is 60, ranging from 0 to 60, the higher the score the worse will be the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hafeez, MBBS, Study Chair — CMH Lahore
Locations (1):
- Cmh Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No